CLINICAL TRIAL: NCT06620055
Title: Development of an Artificial Intelligence Model for Optimising Therapy in Gliomas
Brief Title: Development of an Artificial Intelligence Model for Optimising Therapy in Gliomas Gliomas
Acronym: GLIO-AI
Status: Recruiting | Type: Observational
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Responsible Party: Sponsor
Other Study IDs: CRO-2023-40
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Artificial intelligence (AI) undoubtedly represents the main tool currently available in the definition of complex algorithms and its use in the medical field is becoming increasingly strategic.As reported in the literature, it is increasingly difficult to find new therapeutic strategies for neoplasms, especially neurological ones. Molecular characterisation is therefore increasingly essential, as is the use of new predictive methods.

With this in mind, the aim of this study is to assess, by means of AI algorithms applied to genomic data, in what percentage molecular alterations are susceptible to potential drug therapies, compared to the literature data that does not consider AI algorithms for this purpose.

DETAILED DESCRIPTION:
Artificial intelligence (AI) undoubtedly represents the main tool currently available in the definition of complex algorithms and its use in the medical field is becoming increasingly strategic.As reported in the literature, it is increasingly difficult to find new therapeutic strategies for neoplasms, especially neurological ones. Molecular characterisation is therefore increasingly essential, as is the use of new predictive methods.

With this in mind, the aim of this study is to assess, by means of AI algorithms applied to genomic data, in what percentage molecular alterations are susceptible to potential drug therapies, compared to the literature data that does not consider AI algorithms for this purpose.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a histopathological diagnosis of glioma for whom it is possible to have cryopreserved or fixed in formalin and embedded in paraffin biological material. Specimens may result from incisional biopsy and/or surgical resection and/or blood. Whole blood is taken for germinal analysis;
2. Age >=18 years;
3. Patients must understand and provide written informed consent;
4. Life expectancy >3 months;
5. Presence of biological material from resection and blood considered sufficient by quality and quantity to proceed to molecular characterisation in the opinion of the Investigator Principal Investigator;
6. Presence of available and accessible clinical and histopathological data.

Exclusion Criteria:

1. Refusal of informed consent;
2. Uncooperative patients;
3. Presence of other neoplastic diseases in the last 5 years;
4. Pregnant and/or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 164 patients with a histopathological diagnosis of glioma
Sampling Method: Non-Probability Sample
Enrollment: 164 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2028-11-16 (Estimated); Study Completion 2028-11-16 (Estimated)

PRIMARY OUTCOMES:
proportion of patients, out of total patients number, with molecular characteristics susceptible to potential drug therapies ('druggable') identified using an AI model | 24 months
  proportion of patients, out of total patients number, with molecular characteristics susceptible to potential drug therapies ('druggable') identified using an AI model

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Toffoli, Principal Investigator — Centro di Riferimento Oncologico di Aviano (CRO) - IRCCS; Maurizio Polano, Study Chair — Centro di Riferimento Oncologico di Aviano (CRO) - IRCCS
Locations (3):
- Italy (3):
  - Centro di Riferimento Oncologico (CRO) di Aviano - IRCCS, Aviano, Pordenone
  - IOV, Padua
  - Azienda Sanitaria Universitaria Friuli Centrale (ASUFC, Udine